CLINICAL TRIAL: NCT01268995
Title: A Randomized, Prospective Trial to Evaluate the Effect of Conversion From Tacrolimus to Cyclosporine A After Early Initiation of Insulin Therapy in Patients With New-onset Diabetes Mellitus After Kidney Transplantation
Brief Title: Improving Secretion of Insulin in New Onset Diabetes After Renal Transplantation
Acronym: ISINODAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was impossible to recruit the scheduled number of patients
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Marcus Säemann, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2009-012712-40
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: New Onset Diabetes Mellitus After Renal Transplantation
Keywords: NODAT; kidney transplantation; beta cell function; insulin; Tacrolimus; Cyclosporine A
MeSH Terms: conditions — Insulin Resistance | interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Experimental): Patients in this arm will be switched from immunosuppressive therapy with Tacrolimus to Cyclosporine A. Furthermore, patients in this arm will commence insulin treatment with NPH-insulin to reach normoglycemia. After the achievement of normoglycemia the insulin treatment will be continued for three more weeks and than terminated.
  Interventions: Drug: Cyclosporine A
- Tacrolimus (Active Comparator): Patients in this arm will remain on their immunosuppressive therapy with Tacrolimus. Furthermore, patients in this arm will commence insulin treatment with NPH-insulin to reach normoglycemia. After the achievement of normoglycemia the insulin treatment will be continued for three more weeks and than terminated.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporine A — Patients randomized into arm A will be switched from Tacrolimus to Cyclosporine A. Conversion will be done by a "stop and go" protocol. Patients will take their last dose Tacrolimus in the morning of the day of conversion and will start taking Cyclosporine A in the evening of the same day at a dose of 3mg/kg/d. The first measurement of Cyclosporine A trough levels will be performed 3 days after conversion and the dose will then be adjusted if necessary. Furthermore, treatment with NPH insulin once daily in the morning will be initiated.
  Arms: Cyclosporine A
Drug: Tacrolimus — Patients in arm B will remain on their immunosuppressive therapy with Tacrolimus. Furthermore, treatment with NPH insulin once daily in the morning will be initiated.
  Arms: Tacrolimus

SUMMARY:
New onset diabetes after transplantation (NODAT) is a frequent and feared complication after kidney transplantation and leads to an increase in cardiovascular complications as well as in the rate of graft loss. Very little data exist on how patients in which NODAT has been diagnosed should be treated. It is suspected that Cylosporine A (Sandimmun, TM) is less diabetogenic than Tacrolimus (Prograf, TM). Furthermore, it has been described that early initiation of insulin treatment in Diabetes mellitus type 2 can preserve and improve the function of the insulin secreting cells in the pancreas. Therefore, the investigators test the effects of conversion from Tacrolimus to Cyclosporine A in patients with newly diagnosed NODAT who have just started early treatment with insulin. The hypothesis is that patients who are treated with insulin and who are switched to Cyclosporine A have improved glucose metabolism compared to patients who are treated with insulin and who remain on Tacrolimus therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed NODAT defined by pathologic OGTT (2h, 75mg glucose):

glucose ≥ 200mg/dl

* Defect in insulin secretion as judged by OGTT and HOMA B
* Renal transplantation (deceased or living donor) and treatment with the standard immunosuppression at our center, consisting of tacrolimus, mycophenolate mofetil, prednisone triple therapy without any induction
* stable graft function for more than 3 months post transplant
* informed consent of the patient

Exclusion Criteria:

* patients with prior history of type 1 or type 2 diabetes
* time since transplantation more than 20 years
* allergy against long-acting insulin or cyclosporine A
* body mass index (BMI) > 35
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-09; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
90 days OGTT | 90 days
  The primary endpoint will be the difference in the 2h glucose value obtained from an oral glucose tolerance test (OGTT) after 90 days compared to baseline.

SECONDARY OUTCOMES:
Beta cell function | 90 and 180 days
  One secondary endpoint is the change in beta cell function after 90 days compared to baseline as determined by a frequent sampling oral glucose glucose tolerance test.
Graft rejection | whole study period
  The rate of episodes of acute allograft rejection will be compared between the two treatment arms.
Hypoglycemia | whole study period
  The rate of clinically relevant hypoglycemic episodes will be desribed.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna/General Hospital, Vienna, Austria